CLINICAL TRIAL: NCT02613793
Title: A Prospective Case Control Feasibility Study to Investigate the Utility of Saccadometry in the Diagnosis and Monitoring of Preterm Pre-eclampsia
Brief Title: Saccadic Reaction Time and Preterm Pre-eclampsia
Status: Terminated | Type: Observational
Why Stopped: unable to recruit in suitable time frame
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Lucy MacKillop, Consultant Obstetric Physician, Oxford University Hospitals NHS Trust
Other Study IDs: a11496
Record Dates: First submitted 2015-09-02; First posted 2015-11-25 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Pre-eclampsia
Keywords: Preterm pre-eclampsia; Neurological dysfunction; Saccadic reaction time
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm pre-eclampsia (cases): Pregnant patients diagnosed with pre-eclampsia prior to 35 weeks gestation
- Pregnant patients (controls): Age- and gestation-matched pregnant patients who are not suffering with pre-eclampsia, hypertensive disease or any other neuropsychiatric condition

SUMMARY:
This study is recruiting two groups of women over the age of 18; those who are pregnant and who have pre-eclampsia; and those who are pregnant but do not have pre-eclampsia. The aim is to test a new method of diagnosing and monitoring pre-eclampsia and thus prevent the long-term damage it can cause to the baby's health. Untreated, pre-eclampsia can lead to seizures in pregnancy (eclampsia) and may prove fatal for mother and child.

Currently the only effective treatment for pre-eclampsia is control of the mother's blood pressure until it is safe to deliver the baby. The timing of delivery is kept under constant review by the medical team, who must balance the risk to the mother of developing eclampsia against the risk to the baby of being born too early (premature).

If pre-eclampsia can be diagnosed early, there is a greater chance of being able to treat it effectively. We know that women with pre-eclampsia often have exaggerated reflexes in their limbs (hyperreflexia) and that this may be linked to the risk of seizures. Measuring these reflexes might therefore be a useful way to diagnose and monitor pre-eclampsia, but doing this is not easy, so we want to assess whether measuring other reaction times might similarly help assess the risk of seizures. One possibility is by measuring the reaction time as we flick our eyes to follow a moving target, using an instrument called a saccadometer, which is worn on a head-band, a little like a head-torch.

By comparing the results between these groups and the non-pregnant women, we will be able to see if reaction times from the saccadometer are altered in women with pre-eclampsia, and, if so, whether saccadometry might be useful in helping doctors decide the best time for safe delivery.

DETAILED DESCRIPTION:
Prospective feasibility study with two arms; (i) case-control comparisons of saccadic reaction time distributions between patients with preterm pre-eclampsia, age- and gestation-matched pregnant controls and age-matched female non-pregnant controls [cross-sectional analysis]; (ii) intra-individual comparisons of antenatal and postnatal saccadic reaction time distributions of patients with preterm pre-eclampsia [longitudinal analysis].

ELIGIBILITY:
Inclusion criteria for cases:

1. Age ≥ 18 years
2. Confirmed diagnosis of pre-eclampsia, as defined by the International Society for the Study of Hypertension in Pregnancy (ISSHP)
3. Gestational age < 35+0 weeks
4. Participant is willing and able to give informed consent

Inclusion criteria for controls:

1. Age ≥ 18 years
2. Absence of essential hypertension and pre-eclampsia or pregnancy-induced hypertension in current and previous pregnancies
3. Gestational age < 35+0 weeks
4. Participant is willing and able to give informed consent

Exclusion Criteria:

1. Maternal neurological or psychiatric disorder (e.g. epilepsy, migraine, multiple sclerosis, depression, etc.)
2. Use of medication (other than vitamin supplements [cases and controls] and those for treatment or prevention of pre-eclampsia [cases]) during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients with preterm pre-eclampsia diagnosed earlier than 35 weeks gestation (cases) and healthy age- and gestation-matched pregnant patients (controls)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-01; Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Saccadic reaction times in patients with preterm pre-eclampsia | Baseline (Day 0)
  Attainment of 3000 saccades from women with preterm pre-eclampsia

SECONDARY OUTCOMES:
Comparison of median latency of saccadic reaction time | Baseline (Day 0), twice per week from Day 0 for the duration of hospital stay (which is anticipated to be a maximum 10 weeks from Day 0), and then at Day 1, 5 and 42 postpartum
  Intra-individual and case control comparisons of saccadic reaction time median latency
Comparison of standard deviation of saccadic reaction time median latency | Baseline (Day 0), twice per week from Day 0 for the duration of hospital stay (which is anticipated to be a maximum 10 weeks from Day 0), and then at Day 1, 5 and 42 postpartum
  Intra-individual and case control comparisons of standard deviation of saccadic reaction time median latency
Comparison of standard deviation of early saccadic reaction time median latency | Baseline (Day 0), twice per week from Day 0 for the duration of hospital stay (which is anticipated to be a maximum 10 weeks from Day 0), and then at Day 1, 5 and 42 postpartum
  Intra-individual and case control comparisons of standard deviation of early saccadic reaction time median latency

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Mackillop, BM BCh FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals, Oxford, United Kingdom

REFERENCES:
- [Background] Tuffnell, DJ, Shennan, AH, Waugh, JJS, and Walker, JJ. The management of severe pre-eclampsia/eclampsia, guideline number 10(A). Royal College of Obstetricians and Gynaecologists, London; 2006
- [Background] Irminger-Finger I, Jastrow N, Irion O. Preeclampsia: a danger growing in disguise. Int J Biochem Cell Biol. 2008;40(10):1979-83. doi: 10.1016/j.biocel.2008.04.006. Epub 2008 Apr 11. PMID 18499505
- [Background] Hogberg U. The World Health Report 2005: "make every mother and child count" - including Africans. Scand J Public Health. 2005;33(6):409-11. doi: 10.1080/14034940500217037. No abstract available. PMID 16332605
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Altman D, Carroli G, Duley L, Farrell B, Moodley J, Neilson J, Smith D; Magpie Trial Collaboration Group. Do women with pre-eclampsia, and their babies, benefit from magnesium sulphate? The Magpie Trial: a randomised placebo-controlled trial. Lancet. 2002 Jun 1;359(9321):1877-90. doi: 10.1016/s0140-6736(02)08778-0. PMID 12057549
- [Background] Sibai BM. Management of late preterm and early-term pregnancies complicated by mild gestational hypertension/pre-eclampsia. Semin Perinatol. 2011 Oct;35(5):292-6. doi: 10.1053/j.semperi.2011.05.010. PMID 21962629
- [Background] Liddell E and Sherrington C, Reflexes in Response to Stretch (Myotatic Reflexes. Proceedings of the Royal Society of London. Series B, Containing Papers of a Biological Character, Vol. 96, No. 675 (May 1, 1924), pp. 212-242
- [Background] Carpenter RHS. The saccadic system: a neurological microcosm. Advances in Clinical Neuroscience and Rehabilitation. 2004;4:6-8
- [Background] Hikosaka O, Wurtz RH. Visual and oculomotor functions of monkey substantia nigra pars reticulata. I. Relation of visual and auditory responses to saccades. J Neurophysiol. 1983 May;49(5):1230-53. doi: 10.1152/jn.1983.49.5.1230. No abstract available. PMID 6864248
- [Background] Antoniades CA, Altham PM, Mason SL, Barker RA, Carpenter R. Saccadometry: a new tool for evaluating presymptomatic Huntington patients. Neuroreport. 2007 Jul 16;18(11):1133-6. doi: 10.1097/WNR.0b013e32821c560d. PMID 17589313
- [Background] Michell AW, Xu Z, Fritz D, Lewis SJ, Foltynie T, Williams-Gray CH, Robbins TW, Carpenter RH, Barker RA. Saccadic latency distributions in Parkinson's disease and the effects of L-dopa. Exp Brain Res. 2006 Sep;174(1):7-18. doi: 10.1007/s00221-006-0412-z. Epub 2006 Mar 17. PMID 16544135
- [Background] Chandna A, Chandrasekharan DP, Ramesh AV, Carpenter RH. Altered interictal saccadic reaction time in migraine: a cross-sectional study. Cephalalgia. 2012 Apr;32(6):473-80. doi: 10.1177/0333102412441089. Epub 2012 Apr 5. PMID 22492423
- [Background] Pearson BC, Armitage KR, Horner CW, Carpenter RH. Saccadometry: the possible application of latency distribution measurement for monitoring concussion. Br J Sports Med. 2007 Sep;41(9):610-2. doi: 10.1136/bjsm.2007.036731. Epub 2007 May 11. PMID 17496064
- [Background] Tranquilli AL, Dekker G, Magee L, Roberts J, Sibai BM, Steyn W, Zeeman GG, Brown MA. The classification, diagnosis and management of the hypertensive disorders of pregnancy: A revised statement from the ISSHP. Pregnancy Hypertens. 2014 Apr;4(2):97-104. doi: 10.1016/j.preghy.2014.02.001. Epub 2014 Feb 15. No abstract available. PMID 26104417